CLINICAL TRIAL: NCT01906307
Title: A Phase 1 Study of LJPC-501 in Patients With Hepatorenal Syndrome
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Corporate decision
Sponsor: La Jolla Pharmaceutical Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LJPC-501-CS-5001
Record Dates: First submitted 2013-07-17; First posted 2013-07-24 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2016-03

CONDITIONS: Hepatorenal Syndrome Type I and Type II
Keywords: hepatorenal syndrome
MeSH Terms: conditions — Hepatorenal Syndrome | interventions — Angiotensin I

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LJPC-501 (Experimental): LJPC-501, continuous infusion
  Interventions: Drug: LJPC-501

INTERVENTIONS:
Drug: LJPC-501 — Patients will receive LJPC-501 at titrated doses, with a starting range from 1 to 100 ng/kg/min, by continuous infusion on Days 1 through 5. In Group 1, drug doses will be titrated to 5, 15, and 25 ng/kg/min, after which doses will be titrated in multiples of 25 ng/kg/min. In Groups 2-5, drug doses will be titrated by 25 ng/kg/min. Dose titrations will occur every 2 hours until a MAP of 110 mmHg is reached, maximum urine output is achieved, or a dose of 250 ng/kg/min is achieved. Dosing will then continue at the maximum dose achieved through Day 5.

SUMMARY:
Hepatorenal syndrome (HRS) is a life-threatening condition marked by rapid decline in kidney function in patients with liver cirrhosis or fulminant liver failure. Vasodilation in the gastrointestinal region is largely thought to contribute to the disease. LJPC-501 is a vasoconstrictor that may restore proper circulation and kidney function in patients with HRS.

DETAILED DESCRIPTION:
Vasoconstrictors are considered a promising approach to treat HRS due to the significant vasodilation of the splanchnic circulation that contributes to systemic arterial underfilling and leads to functional decline of the kidney in these patients. Vasoconstrictors currently in use are associated with reduced organ perfusion and have marginal effect on sodium excretion. The vasoconstrictor angiotensin II has been shown to produce significant sodium excretion and urine output in patients with cirrhosis and ascites, supporting its potential utility in the treatment of HRS.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with HRS, as defined by the International Ascites Club [1]:

   * Cirrhosis with ascites
   * Serum creatinine > 1.5 mg/dL
   * No improvement of serum creatinine (decrease to a level of ≤ 1.5 mg/dL) after at least 2 days with diuretic withdrawal and volume expansion with albumin
   * Absence of shock
   * No current or recent treatment with nephrotoxic drugs
   * Absence of parenchymal kidney disease, as indicated by proteinuria > 500 mg/day, microhematuria (> 50 red blood cells per high power field) and/or abnormal renal ultrasonography

   Or patients with HRS due to acute alcoholic hepatitis
2. Patient is able to undergo a reliable neurologic exam, as determined by the investigator
3. Patient or legal surrogate is willing and able to provide written informed consent
4. Patient is willing and able to comply with all protocol requirements

Exclusion Criteria:

1. Evidence of shock
2. Current or recent treatment with nephrotoxic drugs
3. Use of midodrine, octreotide, or other vasopressors within 48 hours of screening
4. Current treatment with dialysis
5. Serum creatinine > 7 mg/dL
6. Active cardiovascular disease within 3 months of screening
7. History of transient ischemic attacks or prior stroke
8. History of organ transplant
9. Ongoing infection requiring intravenous administration of antibiotics (patients with documented infections considered by the Investigator to be controlled within 48 hours of screening may be permitted in the study upon consultation with the Sponsor's Medical Monitor)
10. Participation in a clinical trial within 30 days of screening
11. Patient unlikely to survive more than 72 hours in the opinion of the investigator
12. Patient is pregnant or planning to become pregnant during study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2014-03; Primary Completion 2015-11 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Adverse events through 5 days of treatment | 5 days

SECONDARY OUTCOMES:
Maximum Tolerated Dose | 5 days
Effects on serum creatinine through 5 days of treatment | 5 days
Effects on ascites through 5 days of treatment | 5 days
Effects on urine output through 5 days of treatment | 5 days
Effects on sodium excretion through 5 days of treatment | 5 days

OTHER OUTCOMES:
Change in biomarkers of disease activity from baseline on Day 5 | baseline and Day 5

CONTACTS AND LOCATIONS:
Overall Officials: George Tidmarsh, MD, PhD, Study Director
Locations (1):
- Annette C. & Harold C. Simmons Transplant Institute @ Baylor University Medical Center, Dallas, Texas, United States